CLINICAL TRIAL: NCT05934318
Title: Oral Antenatal L-citrulline Supplementation to Reduce Adverse Pregnancy Outcomes: a Two-arm, Randomized, Placebo-controlled Multi-site Trial in Kenya
Brief Title: L-ArGinine to pRevent advErse prEgnancy Outcomes (AGREE)
Acronym: AGREE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool School of Tropical Medicine (Other)
Collaborators: Kenya Medical Research Institute (Other); University of Toronto (Other); Telethon Kids Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 19-109; PACTR202303697293140 (Registry Identifier: The Pan African Clinical Trials Registry (PACTR))
Record Dates: First submitted 2023-04-05; First posted 2023-07-06 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Pregnancy; Malaria; Nutrition; Placental Development; Preterm Birth; Fetal Growth Restriction
MeSH Terms: conditions — Malaria; Premature Birth; Fetal Growth Retardation | interventions — Citrulline; Arginine

STUDY DESIGN:
Intervention Model Description: * Allocation: randomised; Intervention model: parallel assignment
  * Design: Superiority trial
  * Arms: two
  * Allocation ratio: 1:1; stratified by site (hospital) and gravidity (pauci,- and multigravidae) Masking: placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study will be placebo-controlled involving a maltodextrin/lactose anhydrous/citric acid/lemon flavour powder for the L-citrulline powder intervention. The placebo powder will be indistinguishable in size, quantity, taste and colour from the L-citrulline product to ensure blinding of all investigators and study staff during allocation and for the duration of the trial. All participants and the clinical and research staff will be masked to the treatment assignment of these individual women. The trial statistician will also be blinded regarding the treatment code when s/he develops the statistical analysis plan and writes the statistical programmes, which will be validated and completed using dummy randomisation codes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- L-citrulline arm (Experimental): L-citrulline arm is the intervention arm consisting of a twice daily 6.0 g sachet, each containing 5.000 g of quality-assured L-citrulline powder, 0.672 g maltodextrin and 0.286 g lactose anhydrous, 0.03 g citric acid, 0.012 g lemon flavour + antenatal standard of care with enhanced monitoring. The sachets will be provided at enrolment and each subsequent monthly ANC visit.
  Interventions: Dietary Supplement: L-citrulline
- Placebo arm (No Intervention): Placebo arm is the control arm consisting of a twice daily 6.0 g sachet of quality-assured placebo, each consisting of 3.6 g maltodextrin and 2.358 g lactose monohydrate, 0.03 g citric acid, 0.012 g lemon flavour + antenatal standard of care with enhanced monitoring. The sachets will be provided at enrolment and each subsequent monthly ANC visit.

INTERVENTIONS:
Dietary Supplement: L-citrulline — Twice daily 6.0 g sachet, each containing 5.00 g of quality-assured L-citrulline powder, 0.66 g maltodextrin and 0.30 g lactose anhydrous, 0.03 g citric acid, 0.01 g lemon flavour + antenatal standard of care with enhanced monitoring
  Other Names: L-arginine
  Arms: L-citrulline arm

SUMMARY:
There are few safe, effective, and affordable interventions to improve pregnancy outcomes in low resource settings where the highest rates of poor birth outcomes occur. L-citrulline is naturally found in many foods and is changed into another important amino acid, L-arginine, in the body. L-arginine is important for the growth of a healthy placenta and healthy baby. Adding L-citrulline to the diets of pregnant women may be an effective and affordable way to improve the health of their babies.The goal of the AGREE trial is to test whether a dietary supplement containing a common food component, an amino acid called L-citrulline, can help pregnant Kenyan women at risk of malaria have healthier pregnancies and healthier babies. 2,960 pregnant Kenyan women will be enrolled and randomly assigned to take either a twice daily dietary supplement containing L-citrulline or a placebo supplement without additional L-citrulline. Maternal participants will be seen every month until delivery and at weeks 1 and 6 after birth. Infants will also be followed up at ages 6, 12, 18, and 24 months. The primary outcome of the study is 'adverse pregnancy outcome', a composite of foetal loss (miscarriage or still birth), preterm birth, low birth weight, small for gestational age or neonatal mortality. The results of the AGREE trial could help to guide obstetric and public health policy and provide a sustainable solution that could be implemented at the community level.

DETAILED DESCRIPTION:
L-arginine is an essential amino acid in pregnancy and a key mediator of placental development and function. In many low-resource settings, widespread protein undernutrition contributes to L-arginine deficiency in pregnancy which is associated with an increased risk of adverse pregnancy outcomes. Using a preclinical model, we have previously shown that dietary L-arginine supplementation enhances placental vascular development and improves pregnancy outcomes. L-citrulline is an amino acid that is efficiently converted to L-arginine in the body and has a more palatable flavour profile. The primary objective is to to determine if daily antenatal oral supplementation with L-citrulline can reduce adverse pregnancy outcomes (defined as a composite of fetal loss, infants born preterm, small for gestational age or with low birthweight) among pregnant women at high risk of malaria and protein undernutrition in Kenya.This is an individually randomized, two-arm, parallel-group, placebo-controlled clinical trial involving 2,960 pregnant women randomly assigned to one of two study arms. The intervention arm will contain L-citrulline arm -twice daily 6.0 g sachet, each containing 5.00 g of quality-assured L-citrulline powder, 0.66 g maltodextrin and 0.30 g lactose anhydrous, 0.03 g citric acid, 0.01 g lemon flavour + antenatal standard of care with enhanced monitoring (n=1,480); or placebo arm containing 6.0 g sachet of quality-assured placebo, each consisting of 3.6 g maltodextrin and 2.4 g lactose monohydrate, 0.03 g citric acid, 0.01 g lemon flavour + antenatal standard of care with enhanced monitoring (n=1,480). All participants will continue to take the assigned product for 6 weeks after delivery and will receive an enhanced antenatal standard of care. The primary outcome is the clinical composite 'adverse pregnancy outcome'. Secondary outcomes include longitudinal assessments of physiological and molecular markers of endothelial function, angiogenesis, inflammation, placental function, L-arginine metabolism, neonatal sepsis, mortality, and early childhood neurocognitive development to age 24 months. The effect of L-citrulline supplementation on the composition of the participants' vaginal microbiota and the intestinal microbiota of both the participants and their newborns will be analysed in a subset of 132 mother/infant dyads. All maternal participants of the AGREE trial will be followed for 6 weeks post-partum and the children will be followed until age 2 years. Written informed consent will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged 16-40 years,
* inclusive to 24 weeks gestational age as confirmed by ultrasound,
* who have a viable singleton pregnancy,
* are residents of the study area,
* willing to adhere to scheduled and unscheduled study visit procedures,
* willing to deliver in a study clinic or hospital

Exclusion Criteria:

* multiple pregnancies (i.e. twin/triplets);
* pre-existing hypertension, renal disease and/or diabetes, or severe anaemia (Hb < 5 g/dL);
* HIV-positive or HIV status unknown;
* malformations or nonviable pregnancy observed on enrolment ultrasound;
* known allergy or contraindication to any of the study supplements including lactose intolerance or observing a lactose-free diet;
* unable to give consent; or concurrent participation in any other clinical trial

Ages: 16 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Pregnant women
Enrollment: 2960 (Estimated)
Dates: Start 2023-12-29 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Adverse pregnancy outcome | 27 months
  The primary outcome is 'adverse pregnancy outcome' defined as a composite of fetal loss (spontaneous abortion or stillbirth), singleton live births born SGA or with LBW, or preterm birth (PTB). 'Small for gestational age' will be defined using the INTERGROWTH population reference's 10th percentile. Fetal loss will be assessed monthly at scheduled ANC visits.

SECONDARY OUTCOMES:
Gestational hypertension | 27 months
  Assessed with systolic and diastolic blood pressure
Malaria infection during pregnancy | 27 months
  detected by microscopy and PCR (not for point of care) on peripheral blood
Placental malaria | 27 months
  detected by microscopy, by molecular methods, or by histology (past and active infection) on placental samples
Individual components of the placental malaria composite | 27 months
  detected by microscopy, by molecular methods, or by histology (past and active infection) on placental samples
Uncomplicated clinical malaria during pregnancy | 27 months
  RDTs will be used at the point of care for any patient presenting with fever, history of fever within 48h, or any other symptoms of clinical malaria infection. RDT-positivity is defined as either pLDH or HRP2 antigen positivity.
SARS-CoV-2 infection during pregnancy | 27 months
  Plasma samples will also be assayed for SARS-CoV-2 antibodies using validated techniques available at the time of analysis. If women are symptomatic a rapid SARS-COV-2 antigen test will also be conducted. If the rapid SARS-COV-2 antigen test is negative a confirmatory PCR will be conducted.
Maternal anaemia during pregnancy and delivery | 27 months
  Maternal anaemia is defined as haemoglobin concentration (Hb)<11g/dL; moderate maternal anaemia: Hb<9g/dL); severe anaemia: Hb<7g/dL); congenital anaemia: newborn Hb<12.5 g/dL.
Individual components of the adverse pregnancy outcome composite, and sub-composites | 27 months
  Including fetal loss (spontaneous abortions and stillbirth) and adverse livebirth (SGA-LBW-PTB composite). Gestational age will be assessed using ultrasound dating at enrolment. Preterm birth is defined as <37 weeks' gestation. Newborns will be weighed within 24 hours of delivery using digital scales (± 10 g) with LBW defined as <2,500g. Small for gestational age (SGA) will be defined as birth weight below the tenth percentile for a given gestational age and sex using the new INTERGROWTH reference population. Neonatal length and stunting will be assessed within 24 hours of delivery. Infants will be defined as stunted if their height-for-age is more than two standard deviations below the WHO Child Growth Standards median.
Fetal growth | 27 months
  estimated by validated ultrasound and maternal biomarkers
Birthweight-for-gestational age | 27 months
  Gestational age will be assessed using ultrasound dating at enrolment. Small for gestational age (SGA) will be defined as birth weight below the tenth percentile for a given gestational age and sex using the new INTERGROWTH reference population.
Neonatal length and stunting | 27 months
  Newborns will be measured for length within 24 hours of delivery. Infants will be defined as stunted if their height-for-age is more than two standard deviations below the WHO Child Growth Standards median.
Congenital anaemia | 27 months
  congenital anaemia: newborn Hb<12.5 g/dL.
Congenital malaria infection | 27 months
  detected by microscopy and PCR (not for point of care) on cord blood samples
Congenital SARS-CoV-2 infection | 27 months
  SARS-CoV-2 antibodies detected on cord blood samples
Neonatal death | 27 months
  vital status on discharge (alive/dead), vital status at 7 days (alive/dead) and 28 days (alive /dead) post admission will be documented.
Perinatal mortality | 27 months
  vital status on discharge (alive/dead), vital status at 7 days (alive/dead)
Composite of fetal loss and neonatal mortality | 27 months
  miscarriage, still births or vital status on discharge (alive/dead), vital status at 7 days (alive/dead) and 28 days (alive /dead) post admission will be documented.
Neonatal sepsis | 27 months
  WHO Integrated Management of Childhood Illness criteria128, specifically any one of the following signs (i) not able to feed at all or not feeding well, (ii) convulsions, (iii) severe chest indrawing, (iv) high body temperature (380C or above), (iv) low body temperature (less than 35.50C), (v) movement only when stimulated or no movement at all (vi) in infants less than 7 days old, fast breathing (60 breaths per minute or more).
Early childhood neurocognitive development | 27 months
  Early childhood neurocognitive development will be assessed longitudinally over the first two years of life using a combination of questionnaires, direct assessments, and objective measures appropriate to the developmental periods within this time frame. The Home Observation for Measurement of the Environment (HOME) is a 58-question assessment. The WHO Motor Development Milestones checklist is a simple, WHO-validated assessment of six gross motor milestones in early childhood development. The Mullen Scales of Early Learning (MSEL) is a comprehensive evaluation assessing early childhood development in five domains. The MacArthur Bates Communication Developmental Inventory (MCAB-CDI)132 is an interview-style questionnaire that consists of 100 vocabulary items, 6 gesture items, and 5 grammatical items to assess communication/language development.
Allergic reaction | 27 months
  defined as anaphylaxis, hives/rash after taking the supplement.
Maternal mortality | 27 months
  Maternal mortality will be defined as the death of a woman while pregnant or within 42 days of termination of pregnancy, irrespective of the duration and site of the pregnancy, from any cause related to or aggravated by the pregnancy or its management but not from accidental or incidental causes. A verbal autopsy questionnaire will attempt to determine the cause of death.
Congenital abnormalities | 27 months
  any abnormality detected in surface and clinical examination at birth and week 1 and 6-8
Vomiting study supplement | 27 months
  vomiting within 30 minutes of taking the supplement
Gastrointestinal complaints | 27 months
  including nausea, dyspepsia, diarrhea reported at scheduled and unscheduled visits and and through follow-up phone calls and home visits
Symptoms of dizziness or syncope or palpitations | 27 months
  Study staff will administer a questionnaire to assess for the occurrence of tolerability adverse events (including nausea, dyspepsia, diarrhoea, dizziness, palpitations) at scheduled and unscheduled visits, and and through follow-up phone calls and home visits
Markers of L-arginine bioavailability and nitric oxide biogenesis | 27 months
  L-arginine bioavailability will be assessed by plasma concentrations of L-arginine, ADMA and the L-arginine/ADMA ratio. Plasma SDMA will also be quantified.
Markers of endothelial function, placental function and inflammation | 27 months
  including plasma concentrations of Angiopoietin (Ang)-1, Ang-2, soluble Tyrosine kinase with immunoglobulin-like and EGF-like domains (sTIE)1, sTIE2, Vascular Endothelial Growth Factor (VEGF), soluble VEGF-receptor1, soluble Endoglin (sEng), Placental Growth Factor (PLGF), soluble Intercellular Adhesion Molecule (sICAM), soluble Tumour Necrosis Factor (sTNF) receptor 2 (sTNFR2), C5a, Chitinase-3-like protein 1 (CHI3L1), C-reactive protein (CRP), Interleukin (IL)-18 binding protein (IL-18BP), IL-6, Pregnancy-associated Protein A (PAPP-A), beta-human chorionic gonadotropin (β-hCG); and urine concentrations of protein and complement
Evidence of malaria or SARS-CoV-2 vertical transmission | 27 months
  Laboratory and nutritional outcomes
Evidence of SARS-CoV-2 infection | 27 months
  Laboratory and nutritional outcomes: (antigen, PCR, and/or serology)
Mediators of host immune function | 27 months
  Concentrations of circulating mediators of host immune function, response, endothelial function, and nutrition in the newborn at birth and six weeks of life
Microbial diversity | 27 months
  (N=132 maternal and N=132 newborn participants). Shannon diversity and other measures of microbial diversity richness and abundance in maternal intestinal and vaginal microbiota at enrolment and the first post-treatment timepoint, across gestation and at six weeks post-partum, and in newborn intestinal microbiota at six weeks of life. Nutritional and microbial composition of breast milk

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Kain, PhD, Principal Investigator — University of Toronto; Julie Wright, MD, Study Director — University of Toronto
Locations (1):
- KEMRI Centre for Global Health Research, Kisumu, Kenya

IPD SHARING:
Plan to Share IPD: Yes
Biological samples and data will be shared using material and data transfer agreements with the collaborating institutions to minimise the risk of unauthorised analysis beyond the scope of the agreed parameters. The full protocol will be available on request to any interested professional and may be published in peer-reviewed journals or deposited in an online repository. Individual, de-identified participant data will be made available for meta-analyses as soon as the data analysis is completed, with the understanding that results of the meta-analysis will not be published prior to the results of the individual trial without the prior agreement of the investigators. A fully de-identified data set of the complete patient-level data will be available for sharing purposes, such as via WWARN repository platform http://www.wwarn.org/working-together/sharing-data/accessing-data).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: No later than five years after the publication of the trial.
Access Criteria: Collaborating institutions. All requests for data for secondary analysis will be considered by the Data Access Committee to ensure that the use of data is within the terms of consent and ethics approved.